CLINICAL TRIAL: NCT00688844
Title: Baseline Evaluation and Long-term Follow-up of Nutritional Status and Neurotransmitter Concentrations in Phenylketonuria Patients Initiating Treatment With Sapropterin Dihydrochloride (KuvanTM), a Tetrahydrobiopterin Analog.
Brief Title: Nutritional and Neurotransmitter Changes in PKU Subjects on BH4
Acronym: BH4&PKU
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: BioMarin Pharmaceutical (Industry); Atlanta Clinical and Translational Science Institute (Other)
Responsible Party: Principal Investigator, Rani Singh, Associate Professor, Emory University
Other Study IDs: IRB00007828
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Phenylketonuria
Keywords: PKU; Phenylketonuria; BH4; Kuvan; Tetrahydrobiopterin; Sapropterin Dihydrochloride; Nutrition; PHE; Phenylalanine; PAH; Phenylalanine hydroxylase; Neurotransmitters; Serotonin; Catecholamines; Diet; Body Fat; Bone Density
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma Blood platelets Whole blood Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PKU subjects - baseline: Male and female subjects with PKU at baseline starting KuvanTM therapy.
  Interventions: Drug: KuvanTM Therapy

INTERVENTIONS:
Drug: KuvanTM Therapy — BH4 treatment was prescribed by each participant's medical provider, not an intervention that was assigned as part of the current study.
  Other Names: BH4; Kuvan

SUMMARY:
HYPOTHESIS: The investigators hypothesize that KuvanTM therapy could influence nutritional and body composition parameters and neurotransmitter concentrations in pediatric and adult PKU subjects.

SUMMARY: Though the investigators know that KuvanTM lowers blood Phe levels and improves tolerance for natural protein in at least half of the PKU (Phenylketonuria) patient population, investigators do not know the full effects this medicine will have on the patient's diet, or what impact the medicine or diet changes will have on the body composition or nutrient status of PKU patients. Since KuvanTM may also help the body produce neurotransmitters, investigators also want to find out if taking KuvanTM changes neurotransmitter levels in PKU patients, and if PKU patients who are benefitting from KuvanTM feel less stigmatized and have a better outlook on life as a result of the treatment.

Therefore, the research study has several objectives. These are to investigate the impact KuvanTM therapy has on (1) body composition parameters of PKU patients: such as lean body mass, percent body fat, bone density, weight gain, and growth (2) dietary changes, and the effect of those changes, on intake of calories and essential nutrients (3) changes in blood biomarkers of certain nutrients (4) blood and urine neurotransmitter levels, since these changes could indicate improved neurological functioning, (5) and quality of life of PKU patients, who may feel less burdened due to the dietary freedom KuvanTM provides.

DETAILED DESCRIPTION:
BACKGROUND : Tetrahydrobiopterin (BH4) is a treatment option newly available to phenylketonuria (PKU) patients within the United States as the pharmaceutical KuvanTM. This small molecule functions as a cofactor in multiple enzyme systems, including the metabolism of phenylalanine into tyrosine by the enzyme phenylalanine hydroxylase (PAH).

HYPOTHESIS: The investigators hypothesize that KuvanTM therapy could influence nutritional and body composition parameters and neurotransmitter concentrations in pediatric and adult PKU subjects.

OBJECTIVES:

1. To record nutritional biomarkers, body composition, bone density, and measures of nutrient intake in a phenylketonuria subject group at baseline and for one year after start of KuvanTM therapy.
2. To investigate changes in monoamine neurotransmitter synthesis in a phenylketonuria subject group at baseline and for one year after start of KuvanTM therapy.
3. Evaluate changes in quality of life (QOL) for PKU subjects beginning KuvanTM therapy

METHODOLOGY: Investigators intend to enroll 60 PKU patients, ages 4 to adulthood, who are planning to begin BH4 treatment as prescribed by their medical provider. Patients will be given 4 weeks to demonstrate a response to KuvanTM as determined by a drop in plasma PHE by ≥15%. All patients, regardless of response to KuvanTM, will be allowed to continue in the study. All subjects will be followed for a full 12 months while monitoring nutrient intake, nutritional biomarkers, serotonin and catecholamine levels, and QOL. Two-tailed statistical analysis with α=0.05 will be used to compare results between responders and nonresponders, as well as compare follow-up values with baseline measures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PKU
* ability to provide informed consent (or have legal guardian who can provide informed consent)
* at least 4 years of age
* planning on trying BH4 treatment

Exclusion Criteria:

* Pregnant
* unable to provide informed consent
* less than 4 years of age
* currently taking BH4

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Phenylketonuria (PKU) subjects ages 4 through adulthood who plan to start BH4 therapy but are not currently on BH4.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rani H Singh, PhD, RD, Principal Investigator — Emory University Department of Human Genetics
Locations (2):
- United States (2):
  - Emory Hospital, CIN/ACTSI, Atlanta, Georgia
  - Emory University Genetics Clinic, Decatur, Georgia

REFERENCES:
- [Derived] Jani R, Coakley K, Douglas T, Singh R. Protein intake and physical activity are associated with body composition in individuals with phenylalanine hydroxylase deficiency. Mol Genet Metab. 2017 Jun;121(2):104-110. doi: 10.1016/j.ymgme.2017.04.012. Epub 2017 Apr 28. PMID 28465125
- See also: BH4 & PKU Study Opportunity — http://genetics.emory.edu/research/singh/bh4-pku-study/index.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment lasted 1 year from October 2008 - October 2009. Recruitment occurred at the Emory University Genetics Clinic, Department of Human Genetics in Decatur, GA.
Pre-assignment Details: There were no exclusions of subjects once enrolled.
Groups:
- Subjects With Phenylketonuria Starting Sapropterin Therapy: Subjects with Phenylketonuria starting sapropterin therapy for the purpose of lowering blood phenylalanine levels.
Period: Overall Study
Arm/Group | Subjects With Phenylketonuria Starting Sapropterin Therapy
Started | 58
Completed | 48
Not Completed | 10
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With Phenylketonuria Starting Sapropterin Therapy
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 38
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in BMI at 12 Months
Description: Change in Body mass index (BMI) from baseline of Kuvan study to 12 months post-baseline
Time Frame: Baseline and 12 months
Population: Data missing for 2 participants
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Subjects With Phenylketonuria Starting Sapropterin Therapy
Number analyzed (Participants) | 46
kg/m^2 | -0.65574 (8.060658)
Statistical Analysis 1: Comparison: Subjects With Phenylketonuria Starting Sapropterin Therapy; Objective was to evaluate BMI across one year in PKU patients introduced to sapropterin after baseline. Study was prospective cohort in design; Test type: Superiority or Other; p = 0.692782, t-test, 2 sided; Mean Difference (Final Values) = -0.655574, Standard Deviation 8.060658

2. Primary Outcome: Change From Baseline in Bone Mineral Density (BMD) at 12 Months
Description: Change in bone mineral density (BMD) from baseline of Kuvan study to 12 months post-baseline
Time Frame: Baseline and 12 months
Population: Data missing for 3 participants
Measure: Mean (Standard Deviation); unit: grams/centimeter^2
Arm/Group | Subjects With Phenylketonuria Starting Sapropterin Therapy
Number analyzed (Participants) | 45
grams/centimeter^2 | 0.005401 (0.0243)
Statistical Analysis 1: Comparison: Subjects With Phenylketonuria Starting Sapropterin Therapy; Objective was to evaluate total body bone mineral density (BMD) one year via DXA in PKU patients introduced to sapropterin after baseline. Study was prospective cohort in design; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 0.005401, Standard Deviation 0.0243

3. Primary Outcome: Change From Baseline in Percent (%) Lean Mass at 12 Months
Description: % lean mass was measured via dual energy x-ray absorptiometry (DXA)
Time Frame: Baseline and 12 months
Population: Data missing for 3 participants
Measure: Mean (Standard Deviation); unit: Percent Lean Mass
Arm/Group | Subjects With Phenylketonuria Starting Sapropterin Therapy
Number analyzed (Participants) | 45
Percent Lean Mass | 2.419224 (3.4666)
Statistical Analysis 1: Comparison: Subjects With Phenylketonuria Starting Sapropterin Therapy; Objective was to evaluate % lean mass across one year via DXA in PKU patients introduced to sapropterin after baseline. Study was prospective cohort in design; Test type: Superiority or Other; p = 0.017941, t-test, 2 sided; Mean Difference (Final Values) = 2.419224, Standard Deviation 3.4666

4. Primary Outcome: Change From Baseline in Percent (%) Fat Mass at 12 Months
Description: Percent fat mass measured via dual energy x-ray absorptiometry (DXA)
Time Frame: Baseline and 12 months
Population: Data missing for 3 participants
Measure: Mean (Standard Deviation); unit: Percent Fat Mass
Arm/Group | Subjects With Phenylketonuria Starting Sapropterin Therapy
Number analyzed (Participants) | 45
Percent Fat Mass | 1.208889 (3.519867)
Statistical Analysis 1: Comparison: Subjects With Phenylketonuria Starting Sapropterin Therapy; Objective was to evaluate % fat mass across one year via DXA in PKU patients introduced to sapropterin after baseline. Study was prospective cohort in design; Test type: Superiority or Other; p = 0.026009, t-test, 2 sided; Mean Difference (Final Values) = 1.208889, Standard Deviation 3.51967

5. Primary Outcome: Change From Baseline in Plasma Phenylalanine at 12 Months
Description: Full amino acid panel, including phenylalanine, analyzed in fasting plasma samples.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Subjects With Phenylketonuria Starting Sapropterin Therapy
Number analyzed (Participants) | 48
Micromoles per liter | -67.5187 (362.9412)
Statistical Analysis 1: Comparison: Subjects With Phenylketonuria Starting Sapropterin Therapy; Objective was to evaluate plasma phenylalanine across one year in PKU patients introduced to sapropterin after baseline. Study was prospective cohort in design; Test type: Superiority or Other; p = 0.303864, t-test, 2 sided; Mean Difference (Final Values) = -67.5187, Standard Deviation 362.9412

6. Primary Outcome: Change From Baseline in Total Dietary Protein Intake at 12 Months
Description: Total dietary protein intake assessed through 3-day food records - calculated as average protein intake (grams/day) in the 3 days recorded
Time Frame: Baseline and 12 months
Population: Dietary intake not submitted by 11 participants at 12 months.
Measure: Mean (Standard Deviation); unit: grams per day
Arm/Group | Subjects With Phenylketonuria Starting Sapropterin Therapy
Number analyzed (Participants) | 37
grams per day | -10.9549 (20.10814)
Statistical Analysis 1: Comparison: Subjects With Phenylketonuria Starting Sapropterin Therapy; Objective was to evaluate protein intake (grams per day) across one year in PKU patients introduced to sapropterin after baseline. Study was prospective cohort in design; Test type: Superiority or Other; p = 0.00088, t-test, 2 sided; Mean Difference (Final Values) = -10.9549, Standard Deviation 20.10814

7. Primary Outcome: Change From Baseline in Phenylalanine Intake at 12 Months
Description: Total dietary phenylalanine assessed through 3-day food records - calculated as average phenylalanine intake (grams/day) in the 3 days recorded
Time Frame: Baseline and 12 months
Population: Dietary intake not submitted by 11 participants at 12 months.
Measure: Mean (Standard Deviation); unit: grams per day
Arm/Group | Subjects With Phenylketonuria Starting Sapropterin Therapy
Number analyzed (Participants) | 37
grams per day | 0.131676 (0.797247)
Statistical Analysis 1: Comparison: Subjects With Phenylketonuria Starting Sapropterin Therapy; Objective was to evaluate dietary phenylalanine intake across one year in PKU patients introduced to sapropterin after baseline. Study was prospective cohort in design; Test type: Superiority or Other; p = 0.3811, t-test, 2 sided; Mean Difference (Final Values) = 0.131676, Standard Deviation 0.797247

8. Other Pre Specified Outcome: Change From Baseline in Serotonin at 12 Months
Description: Objective: 1 year prospective cohort of PKU patients introduced to sapropterin (Kuvan)to evaluate peripheral neurotransmitter changes across time.
Time Frame: Baseline and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Subjects With Phenylketonuria Starting Sapropterin Therapy
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 20/58
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Phenylketonuria Starting Sapropterin Therapy (N=58)
Sinus and general respiratory infections (Infections and infestations) | 11 (13) — Patients were asked to keep record of illnesses and other adverse events between visits. Patients were encouraged to call in adverse events that occurred between visits but were also queried at each study visit.
Headache (Nervous system disorders) | 8 (9) — Headaches or migraines reported by patients
Gastrointestinal upset (not flu) (Gastrointestinal disorders) | 3 (3) — Diarrhea or acid reflux
Urinary tract infection (Renal and urinary disorders) | 3 (3) — One UTI case due to congenital kidney deformity which patient had surgically corrected a few weeks later.
Flu and flu-type sickness (Infections and infestations) | 7 (8) — Confirmed and suspected flu as reported by patients
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (6) — Includes sore throat from strep, flu, cold, or general sore throat.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes